CLINICAL TRIAL: NCT06609356
Title: Cardiometabolic Benefit of Reducing Iatrogenic Hyperinsulinemia Using Insulin Adjunctive Therapy in Type 1 Diabetes
Acronym: ACT T1D
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Daniel Moore, Associate Professor of Pediatrics, Division of Pediatric Endocrinology and Diabetes, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 240996
Record Dates: First submitted 2024-09-20; First posted 2024-09-24 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Type 1 Diabetes Mellitus; Glucokinase-Maturity Onset Diabetes of the Young (GCK-MODY); MODY2 Diabetes; Healthy Volunteer
Keywords: type 1 diabetes mellitus; with Glucokinase-Maturity Onset Diabetes of the Young (GCK-MODY); nitric oxide; sodium-glucose cotransporter-2 inhibitors (SGLT2i); healthy volunteer; insulin sensitivity; flow-mediated vasodilation (FMD)
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- High insulin (Experimental): Participants will receive a "high insulin infusion" (Hi-Ins) prior to quantifying insulin resistance and endothelial function. This infusion will result in participants having insulin levels similar to patients with type 1 diabetes for five hours.
  Interventions: Procedure: Study Visit 1; Drug: Placebo; Procedure: Study Visit 2
- Normal insulin (Active Comparator): Participants will receive a "normal insulin infusion" (Eu-Ins) prior to quantifying insulin resistance and endothelial function. This infusion will result in participants having insulin levels similar to people without diabetes and people with GCK-MODY for five hours.
  Interventions: Procedure: Study Visit 1; Drug: Placebo; Procedure: Study Visit 2; Drug: Sodium Glucose Co-transporter 2 (SGLT2) Inhibitor

INTERVENTIONS:
Procedure: Study Visit 1 — Hyperinsulinemic, euglycemic clamp and flow-mediated dilation (FMD) study. The study will randomize participants to first receive a five-hour intravenous insulin infusion to achieve normal plasma insulin concentrations (Eu-Ins) or higher plasma insulin concentrations (Hi-Ins)
Drug: Placebo — * T1DM participants in the Hi-Ins study will receive an oral placebo. During the Eu-Ins study they will receive an SGLT2i.
  * CGK-MODY participants and healthy volunteers will receive placebo in both studies.
Procedure: Study Visit 2 — Hyperinsulinemic, euglycemic clamp and flow-mediated dilation (FMD) study. Insulin levels infused during the five-hour insulin infusion will be opposite of the first visit.
Drug: Sodium Glucose Co-transporter 2 (SGLT2) Inhibitor — Concurrent with starting the five-hour infusion, T1DM participants in the Eu-Ins study will receive an SGLT2i dose (empagliflozin 25 mg).
  Arms: Normal insulin

SUMMARY:
This study aims to understand the heart and blood sugar health benefits of using an adjunctive therapy to lower high insulin levels in people with type 1 diabetes. The investigators will also look at people with a specific type of diabetes called Glucokinase-Maturity Onset Diabetes of the Young (GCK-MODY) and those without diabetes to help interpret the results. The investigators will use a medication that helps the body get rid of sugar, called and SGLT2 inhibitor, with the goal to reduce the body's insulin requirements. The investigators believe this could lead to better heart and blood sugar health, including a better response to insulin and more available nitric oxide, a gas that helps blood vessels function well. The investigators will compare heart and blood sugar health risk factors in participants with type 1 diabetes, participants with Glucokinase-Maturity Onset Diabetes of the Young (GCK-MODY), and non-diabetic healthy volunteers under two conditions: high insulin levels typical of type 1 diabetes and normal insulin levels typical of the other two groups.

ELIGIBILITY:
Inclusion Criteria:

Age: 18-60 years BMI: 18-28 kg/m² Weight: ≥ 50 kg

T1DM Participants:

Duration of T1DM: 1-30 years HbA1c: 5.7-7.5% Insulin Therapy: Using automated insulin delivery

GCK-MODY Participants:

HbA1c: 5.7-7.5% Genetic Confirmation: Positive GCK sequencing

Control Participants:

HbA1c: less than 5.5%

** Exclusion Criteria: Severe Hypoglycemia: ≥1 episode in the past 3 months

Comorbidities:

* Any hospital admissions for diabetic ketoacidosis in the past 6 months
* SBP greater than 140 mmHg and DBP greater than 100 mmHg
* eGFR by MDRD equation of less than 60 mL/min/1.73 m²
* AST or ALT greater than 2.5 times ULN
* Hct less than 35%

Medications:

* Any antioxidant vitamin supplement within 2 weeks before the study
* Any systemic glucocorticoid
* Antipsychotics
* Atenolol, Metoprolol, Propranolol
* Niacin
* Any thiazide diuretic
* Any oral contraceptive pill with greater than 35 mcg ethinyl estradiol
* Growth hormone
* Any immunosuppressant
* Antihypertensive
* Any antihyperlipidemic

Other:

* Pregnancy
* Tanner stage less than 5
* Peri- or post-menopausal women
* Active smoker

T1DM Participants:

Medications: Any diabetes medication except insulin C-peptide: greater than 0.7 ng/mL (fasting)

GCK-MODY Participants:

None specific

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Estimated)
Dates: Start 2025-07-03 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Aim 1: Tissue glucose disposal (TGD) | 8 hours
  The primary outcome will be the difference in tissue glucose disposal (TGD) during a hyperinsulinemic, euglycemic clamp between Eu-Ins and Hi-Ins studies.
Aim 2: Nitric Oxide (NO) bioavailability | 8 hours
  This study aims to determine the difference in hyperinsulinemia-mediated suppression of nitric oxide (NO) bioavailability between Eu-Ins and Hi-Ins studies, as measured by flow mediated dilation (FMD) of the brachial artery.

SECONDARY OUTCOMES:
Secondary outcome for Aim 1: Differences in endogenous glucose production | 8 hours
  This study aims to determine the difference in endogenous glucose production at the end of euinsulinemic vs. hyperinsulinemic infusions
Secondary outcome for Aim 2: Nitroglycerin mediated vasodilation of the brachial artery | 8 hours
  Through the use of flow mediated dilation (FMD), the study aims to determine nitroglycerin mediated vasodilation of the brachial artery.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Moore, MD, PhD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in a published article after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, ICF